CLINICAL TRIAL: NCT00994630
Title: Biomarkers for Bipolar Disorder: Chaperones and Reticulum Endoplasmatic Stress Response CHAP´s Study
Acronym: CHAPS
Status: Suspended | Type: Observational
Why Stopped: fail to get funding
Sponsor: University of Sao Paulo (Other)
Responsible Party: Ricardo Alberto Moreno, University of Sao Paulo
Other Study IDs: CHAPS STUDY
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-05

CONDITIONS: Bipolar Disease Type I

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dna and Rna analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- BP I patients manic phase

SUMMARY:
The purpose of this study is to determine expression of chaperones proteins from the endoplasmatic reticulum stress response system in bipolar I patients (manic phase) compared to healthy controls.

Hypothesis: There is no difference in chaperones proteins expression between bipolar I manic patients and healthy controls

ELIGIBILITY:
Inclusion Criteria:

* Bipolar Disease type I manic phase
* YMRS > 14
* HDRS < 9

Exclusion Criteria:

* Use of lithium, divalproate, or carbamazepine in therapeutic levels over the past 30 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Bipolar Disease type I manic phase
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Moreno, MD, PhD, Principal Investigator — Mood Disorders Program, Institute of Psychiatry, Faculty of Medicine, University of Sao Paulo, Brazil; Marcio G Soeiro de Souza, MD, Study Director — Mood Disorders Program, Institute of Psychiatry, Faculty of Medicine, University of Sao Paulo, Brazil
Locations (1):
- Mood Disorders Program, Institute of Psychiatry, Faculty of Medicine, University of Sao Paulo, São Paulo, São Paulo, Brazil